CLINICAL TRIAL: NCT03008850
Title: Shivering Prevention During Cesarean Section by Intrathecal Injection of Magnesium Sulfate
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MOHAMED F. MOSTAFA, Lecturer of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Shivering, MgSO4
Record Dates: First submitted 2016-12-27; First posted 2017-01-04 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Cesarean Section; Shivering
Keywords: Shivering; Intrathecal; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group M (Active Comparator): 2 ml (10 mg) of 0.5% heavy bupivacaine plus 0.5 ml (25 mg) MgSO4 will be injected intrathecally
  Interventions: Drug: MgSo4
- Group P (Active Comparator): 2 ml (10 mg) of 0.5% heavy bupivacaine plus 0.5 ml normal saline will be injected intrathecally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MgSo4 — Patients will be randomly allocated to one of two groups:
  Group (M): 2 ml (10 mg) of 0.5% heavy bupivacaine plus 0.5 ml (25 mg) MgSO4 will be injected intrathecally.
  Group(P): 2 ml (10 mg) of 0.5% heavy bupivacaine plus 0.5 ml normal saline will be injected intrathecally.
  Arms: Group M
Drug: Placebo — Patients will be randomly allocated to one of two groups:
  Group (M): 2 ml (10 mg) of 0.5% heavy bupivacaine plus 0.5 ml (25 mg) MgSO4 will be injected intrathecally.
  Group(P): 2 ml (10 mg) of 0.5% heavy bupivacaine plus 0.5 ml normal saline will be injected intrathecally.
  Arms: Group P

SUMMARY:
Shivering is a common post-anesthetic complication occurring in up to 65% of patients undergoing spinal or epidural anesthesia. Shivering may interfere with electrocardiogram, blood pressure and oxygen saturation monitoring. In addition, shivering increases oxygen consumption, carbon dioxide production and metabolic rate by up to 400%. Thus, it may result in problems in patients with low cardiac and pulmonary reserves. Preventing shivering could therefore result in better postoperative outcomes or reduce the incidence of post-surgical complications.

DETAILED DESCRIPTION:
Magnesium sulfate (MgSO4) has anti-shivering effects. Moreover, it has potential neuroprotective effects and may enhance neuroprotection against the effects of hypothermia. Intrathecal MgSO4 administration provides effective perioperative analgesia and can prolong the period of anesthesia and sensory blockade without any additional side-effects. However, most of the research on the role of MgSO4 in the prevention of shivering has focused on intravenous infusion of this drug. Few clinical trials have examined the effect of adding intrathecal MgSO4 to anesthetic agents such as bupivacaine to suppress anesthesia-related shivering in patients. Similar to infusion studies, we hypothesized that the addition of intrathecal injection of MgSO4 to bupivacaine would improve perioperative shivering in female patients undergoing elective caesarean section. Few previous studies evaluated neuroaxial anti-shivering effects of intrathecal magnesium and none evaluated the anti-shivering effect of intrathecal MgSO4. Therefore, we elected to use the lowest dosage (25 mg MgSO4) that was formerly utilized for investigation of analgesic effects.

Magnesium sulphate is an intracellular cation with various physiologic functions such as enzyme activation, nerve signal conduction, protein synthesis and vasomotor tonicity regulation. Magnesium sulphate has been used in various clinical situations including preeclampsia, tocolysis, arrhythmias, myocardial ischemia, bronchial asthma and postoperative shivering.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 35years.
2. Undergo elective cesarean section under spinal anesthesia.
3. ASA physical status I-II.
4. Singleton pregnancy.
5. At least 38 weeks gestation.

Exclusion Criteria:

1. Women with history of cardiac, liver or kidney diseases.
2. Women with allergy to amide local anesthetics or medication included in the study.
3. Women with any neurological problem.
4. Any contraindication of regional anesthesia.
5. Failed or insatisfactory spinal block.
6. Preoperative temperature more than 38⁰ C.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Shivering Score | 2 hours
  shivering will be recorded in the recovery room for 2 hours

SECONDARY OUTCOMES:
Visual Analogue Pain Score | 2 hours
  analgesics will be given if visual analogue score ≥ 4
Complications | 2 hours
  percentage of patients with any complications will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Zain E. Hassan, MD, Study Chair — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided